CLINICAL TRIAL: NCT04990635
Title: Investigation of the Correlation of Block Success With Perfusion Index Measurement in Pediatric Surgery Performed Under Caudal Epidural Block Anesthesia"
Brief Title: Evaluation of Caudal Block Success With Perfusion Index
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: MEHMET DURAN (Other)
Collaborators: CDemirci (Unknown)
Responsible Party: Sponsor-Investigator, MEHMET DURAN, MDURAN, Adiyaman University
Organization: Adiyaman University (Other)
Other Study IDs: 2020/8-25
Record Dates: First submitted 2021-07-27; First posted 2021-08-04 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Https://Meshb.Nlm.Nih.Gov/Record/ui?ui=D000081282
Keywords: PERFUSION INDEX, PEDIATRIC CAUDAL BLOCK

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Caudal epidural anesthesia was reported as the first epidural anesthesia technique in 1933, but its use started to become widespread after the 1960s(1). The procedure is safe, easy to apply, has a low incidence of complications, and the total complication rate is 1.5/1000; serious complications are 1/40000 (2,3). There are many methods to demonstrate the success of caudal epidural block. Some of the usual traditional methods are changes in mean arterial pressure, heart rate and cremasteric reflex. These methods are sometimes not objective, but take time. In this study, we will examine whether the success of the block in pediatric patients who underwent caudal epidural block, which is applied in our hospital, is correlated with the success of the block, measured with the finger probe, other than traditional methods, and whether the perfusion index shows faster block success than other traditional methods.

DETAILED DESCRIPTION:
A successful caudal epidural block can provide safe, effective regional anesthesia(4). The overall failure rate of caudal epidural block in pediatric patients is approximately 4% according to the anatomical and developmental abnormalities of the caudal canal(1,5). Therefore, reliable and rapid evaluation of a successful caudal epidural block is important to optimize anesthesia management in pediatric patients. Evaluating the success of the caudal epidural block with traditional methods such as mean arterial pressure(MAP), heart rate and cremaster reflex is completely objective.

The aim of this study is to evaluate whether it will detect the success of caudal epidural block faster than other traditional methods in pediatric patients who underwent surgery with caudal epidural block, using perfusion index values measured with a finger probe.

This research; It is a prospective observational study. In our pediatric patients who routinely underwent caudal epidural block under sedation in our hospital, perfusion index values will be recorded by attaching a probe to the big toe. Perfusion index(PI) is a numerical value for the ratio between pulsatile and non-pulsatile blood flow.(6) PI works by measuring the changes in finger peripheral perfusion through pulse oximetry.(7) If the procedure is successful in patients who underwent caudal epidural block, there is an increase in perfusion in the lower extremities due to sympathetic nerve blockade. Therefore, in our study, we will observe whether perfusion increases by measuring the perfusion index value measured using a finger probe, by attaching the probe to the big toe, before the caudal epidural block is performed and at the 1,5, 7, 10, 15 and 20 minutes after the caudal epidural block. Simultaneously, the mean arterial pressure, heart rate and changes will be recorded by looking at the cremaster reflex in male patients. The finding that shows the presence of the cremaster reflex is to hit the upper inner part of the thigh and to pull the scrotum and testis on the same side. A 15% decrease in pulse rate and an increase in the perfusion index value indicate a successful caudal epidural block. We will examine whether the increase in the perfusion index after these procedures is correlated with the success of the block, and whether the perfusion index shows a faster block success than other traditional methods.

ELIGIBILITY:
Inclusion Criteria:

* lower abdomen/urogenital/lower extremity surgery
* PEDIATRIC GROUP BETWEEN 1-6 YEARS
* Patients with ASA1-2

Exclusion Criteria:

* Neuromuscular disease
* PATIENTS WITH ASA3-4
* Patients with cerebral palsy
* Patients with mental retardation
* Patients with hematological disorders
* Infection in the region to be caudal block

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: PATIENT GROUP BETWEEN 1 YEARS OLD AND 6 YEARS OLD WITH INGUINAL HERNI, HYPOSPADIAS, NON-DESCENDED TESTIC SURGERY
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2021-08-17 (Estimated); Primary Completion 2021-08-18 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
DISPLAYING CAUDAL BLOCK SUCCESS BY PERFUSION INDEX IN PEDIATRIC PATIENT GROUP | PATIENTS PIERFUSION INDEX, PULSE AND TENSION MEASUREMENTS 1.5,7,10,15,20 MINUTES AFTER THE CAUDAL BLOCK IS MADE
  CORRELATION OF CAUDAL BLOCK SUCCESS WITH PERFUSION INDEX VALUE WILL BE EVALUATED APPLICABLE TO SEDATATIZED PEDIATRIC PATIENTS IN LOWER ABONE SURGERIES

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman University, Adıyaman, Turkey (Türkiye)

REFERENCES:
- [Background] Silvani P, Camporesi A, Agostino MR, Salvo I. Caudal anesthesia in pediatrics: an update. Minerva Anestesiol. 2006 Jun;72(6):453-9. PMID 16682915
- [Background] Markakis DA. Regional anesthesia in pediatrics. Anesthesiol Clin North Am. 2000 Jun;18(2):355-81, vii. doi: 10.1016/s0889-8537(05)70168-1. PMID 10935015
- [Background] Sanders JC. Paediatric regional anaesthesia, a survey of practice in the United Kingdom. Br J Anaesth. 2002 Nov;89(5):707-10. PMID 12393767
- [Background] Seyedhejazi M, Taheri R, Ghojazadeh M. The evaluation of upper leg traction in lateral position for pediatric caudal block. Saudi J Anaesth. 2011 Jul;5(3):248-51. doi: 10.4103/1658-354X.84096. PMID 21957401
- [Background] Dalens B, Hasnaoui A. Caudal anesthesia in pediatric surgery: success rate and adverse effects in 750 consecutive patients. Anesth Analg. 1989 Feb;68(2):83-9. PMID 2913854
- [Background] Goldman JM, Petterson MT, Kopotic RJ, Barker SJ. Masimo signal extraction pulse oximetry. J Clin Monit Comput. 2000;16(7):475-83. doi: 10.1023/a:1011493521730. PMID 12580205
- [Background] Huang HS, Chu CL, Tsai CT, Wu CK, Lai LP, Yeh HM. Perfusion index derived from a pulse oximeter can detect changes in peripheral microcirculation during uretero-renal-scopy stone manipulation (URS-SM). PLoS One. 2014 Dec 26;9(12):e115743. doi: 10.1371/journal.pone.0115743. eCollection 2014. PMID 25542000